CLINICAL TRIAL: NCT00333957
Title: Capsule Endoscopy in Cystic Fibrosis-Screening for Small Bowel Disease in Cystic Fibrosis Patient.
Brief Title: Capsule Endoscopy in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: will001-HMO-CTIL
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2007-10

CONDITIONS: Cystic Fibrosis
Keywords: capsule endoscopy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Cystic Fibrosis patients continue to have bowel problems even after adequate pancreatic enzyme supplementation. There may be pathology of the lining of the bowel. Capsule endoscopy will be used to photograph the entire bowel.

DETAILED DESCRIPTION:
The capsule endoscope system (Given Imaging, Ltd.) consists of 3 elements: a disposable capsule (PillCamTM SB) that acquires video images during natural propulsion through the digestive system.

The video-capsule PillCamTM SB has been cleared by the FDA for use in patients over 10 years of age for the detection of small intestinal disorders. It has been used in patients under age 10 and has been placed with the use of a gastroscope in patients unable to swallow the capsule. In fact, a new delivery device has been introduced recently that facilitates placement of the video-capsule in pediatric patients.For the purposes of this study, only patients over age 10 years who are able to swallow the capsule would be enrolled.

There are approximately 450 CF patients in the registry in Israel, with about 300 above the age of 10. Study subjects would be enrolled from this registry population and would be screened for the presence of the contraindications noted above. Patients would be assessed for symptoms of possible small bowel lesions at the time of enrollment including gastrointestinal bleeding, palpable abdominal mass, weight loss, diarrhea, and abdominal pain. Markers of inflammation including stool calprotectin will be assessed in all patients. These data would be recorded for further analysis.

Page

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria would include those subjects with known CF who are able to give informed consent to undergo capsule endoscopy and whose guardians provide consent as well, if applicable. -

Exclusion Criteria

Subjects would be excluded if they were felt to be poor surgical candidates as patients may need to undergo surgery in the rare event of retention of the capsule. Patients genotype and lung function will be noted; patients will be excluded if FEV1 < 40%.

-

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-07; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
We will examine the entire small bowel
of CF opatients

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wilschanski, MBBS, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel